CLINICAL TRIAL: NCT06971614
Title: An Open-Label, International, Multicenter Phase II Study to Evaluate the Efficacy and Safety of Intravesical T3011 Injection in Participants With BCG-Unresponsive High-Risk Non-Muscle-Invasive Bladder Cancer (NMIBC) or BCG-Exposed, Chemotherapy-Unresponsive Intermediate /High-Risk NMIBC
Brief Title: A Study of T3011 in Patients With BCG-Unresponsive NMIBC or BCG-Exposed, Chemotherapy-Unresponsive NMIBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmVira Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVR-T3011-006
Record Dates: First submitted 2025-04-27; First posted 2025-05-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Nonmuscle-invasive Bladder Cancer
Keywords: Nonmuscle-invasive Bladder Cancer; Herpes Virus T3011 Injection; BCG-Unresponsive; BCG-Exposed; Chemotherapy-Unresponsive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T3011 (Experimental): T3011 will be given once a week (QW) for 6 weeks during the induction treatment course, the following 6 weeks are only for observation and then the 3-month efficacy assessment will be conducted. During the maintenance period, T3011 will be given every 3 weeks (Q3W) until about 24 months or meeting the criteria for treatment discontinuation.
  Interventions: Biological: T3011

INTERVENTIONS:
Biological: T3011 — T3011 will be administered at a dose of 1x10^10 PFU intravesically.

SUMMARY:
This is a Phase II clinical study to evaluate the efficacy and safety of intravesical T3011 injection in participants with BCG-unresponsive high-risk NMIBC or BCG-exposed, chemotherapy-unresponsive intermediate/high-risk NMIBC.

DETAILED DESCRIPTION:
In Cohort A, participants will be enrolled with pathologically confirmed high-risk non-muscle invasive bladder cancer (NMIBC) (CIS with or without Ta or T1 papillary) which is unresponsive to BCG treatment.

In Cohort B, participants will be enrolled with pathologically confirmed high-risk non-muscle invasive bladder cancer (NMIBC) (Ta/T1 papillary without CIS) which is unresponsive to BCG treatment.

In Cohort C, participants will be enrolled with pathologically confirmed high-risk non-muscle invasive bladder cancer (NMIBC) (CIS with or without Ta or T1 papillary) which has previously been exposed to BCG and is unresponsive to chemotherapy treatment.

In Cohort D, participants will be enrolled with pathologically confirmed intermediate/high-risk non-muscle invasive bladder cancer (NMIBC) (Ta/T1 papillary without CIS) which has previously been exposed to BCG and is unresponsive to chemotherapy treatment.

In all cohorts, study treatment will be administered as a weekly induction course for the first 6 weeks.

For high-risk participants, a reinduction course administered to participants who have residual CIS or high-grade Ta disease at the 3-month evaluation. Following induction, If the tumor assessment indicates CR or no recurrence the participant enters the maintenance phase, T3011 is administered once every 3 weeks (Q3W).

For intermediate-risk participants, a reinduction course administered to participants who have low-grade Ta disease at the 3-month evaluation. Following induction, the participant achieving no recurrence (e.g., no tumor) enters the maintenance phase, T3011 is administered once every 3 weeks (Q3W).

Disease status will be assessed using cystoscopy, urine cytology, histopathology (if performed), and imaging examinations (if performed) every 3 months during treatment period or until disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

Participants may enter the study only if they meet all the following criteria:

1. Male or female, aged ≥18 years at the time of signing the ICF.
2. The participants will need to meet the following criteria:

   1. Participants with a histologically confirmed diagnosis of NMIBC (Ta, T1 and/or Cis).
   2. During the study, the participants must voluntarily comply with the study-specified cystoscopy, urine cytology and randomized biopsy.
3. All toxicities caused by prior radiotherapy, chemotherapy or other treatments have recovered to Grade ≤1 (CTCAE 5.0) (except for alopecia), including but not limited to urinary tract infection, urinary tract irritation, and macroscopic hematuria; participants with Grade >1 anti-neoplastic treatment-related toxicities during the screening period may be enrolled after discussion of the investigators and the sponsor.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
5. Expected survival ≥24 weeks.
6. Laboratory test values meeting the following requirements :

   1. Hematology ANC≥1.5×10^9/L. PLT count ≥75×10^9/L. Hemoglobin (HGB) ≥90 g/L.
   2. Renal function Creatinine clearance ≥60 mL/min (based on Cockcroft-Gault equation for calculation)
   3. Hepatic function Serum total bilirubin (TBIL) ≤1.5×ULN. Asparate aminotransferase (AST) and alanine transaminase (ALT) ≤2.5×ULN Serum ALB ≥30 g/L.
   4. Coagulation function International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN. Activated partial thromboplastin time (aPTT) ≤1.5×ULN.
7. For women of childbearing potential (WOCBP), the serum pregnancy test prior to the first dose must be negative and the potential participant must promise to use medically acceptable and effective methods of contraception. after signing the ICF until at least 6 months after the last dose.
8. Male participants of child-bearing potential must agree to use medically acceptable and effective methods of contraception after signing the ICF until at least 6 months after the last dose; in addition, male potential participants must agree not to donate sperm during this period.
9. Participants who understand and voluntarily sign the written ICF and are willing and able to comply with all trial requirements.

Exclusion Criteria:

Participants meeting any of the following criteria will not be allowed to participate in this study:

1. Participants meet the following criteria:

   1. Concurrent or prior history of muscle-invasive (muscularis propria) or metastatic bladder cancer.
   2. Urothelial carcinoma of the upper genitourinary tract or prostatic urethra within 24 months prior to investigational product.
   3. Having received chemotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy, investigational product or other anti-neoplastic therapies within 4 weeks prior to investigational product.
   4. Having received radiotherapy within 2 weeks prior to investigational product.
2. Planning to receive any anti-neoplastic therapy other than the investigational products during this study.
3. A history of allergic reactions to HSV-1, IL-12, or anti-PD-1 antibodies or biological components similar to them, or known allergic reactions to any component of the T3011 formulation.
4. A history of brain metastasis or imaging-confirmed brain metastasis , leptomeningeal disease, or spinal cord compression.
5. Concurrent or prior history of other malignancies than that treated in this study.
6. History or evidence of high-risk cardiovascular diseases, including but not limited to:

   1. Serious cardiac rhythm or conduction abnormalities.
   2. Acute myocardial infarction, unstable angina, or stroke, etc., developing within 6 months prior to the first dose of the investigational products.
   3. Coronary angioplasty or stenting within 6 months prior to the first dose of the investigational products.
   4. New York Heart Association (NYHA) criteria-defined cardiac function > Class II; echocardiogram-documented cardiac valve morphological abnormalities (Grade ≥2).
   5. Left ventricular ejection fraction (LVEF) ˂lower limit of normal (LLN) of the study site, or ˂ 50% if no LLN is set at the site.
   6. Poorly controlled blood pressure .
7. The following prior or concurrent immune disorders that in the investigator's opinion would pose unpredictable risks to the participants:

   1. Immune-related pneumonia or other immune-related adverse reactions of Grade ≥3 developing with prior immunotherapy (including but not limited to PD-1/PD-L1).
   2. Concurrent active immune diseases requiring treatment with systemic immunosuppressants (excluding autoimmune diseases not requiring intervention such as vitiligo and diseases treatable by other alternative drugs such as hypothyroidism that is treated with thyroid hormone replacement therapy originally), or concurrent immune diseases requiring treatment with systemic immunosuppressants that have the potential to recurrence (e.g., systemic lupus erythematosus).
   3. Other concurrent diseases require treatment with systemic immunosuppressants.
8. Unexplainable fever >38.5℃ during the screening or on the day of treatment (fever judged as tumor-induced by the investigator is eligible for enrollment) that in the investigator's opinion will affect the participation in this trial or interfere with the efficacy assessment.
9. The following persistent or active infections: human immunodeficiency virus (HIV) antibody-positive, hepatitis B surface antigen [HBsAg] positive with HBV DNA level ≥2000 IU/mL, hepatitis C virus (HCV) antibody positive with detectable HCV RNA, and other active infections requiring systemic treatment.
10. Prior history of splenectomy or organ transplantation.
11. Having previously received treatment with oncolytic virus (e.g., T-VEC, CG0070).
12. Requiring oral or intravenous use of anti-herpes virus drugs, including but not limited to acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscarnet, and cidofovir (except for those to be used locally, such as topically), during the study.
13. Participants with known psychiatric disorders that may affect compliance in trial or with poor compliance.
14. Participants with a history of drug abuse (including "recreational use") or substance abuse (including alcohol) within one year prior to signing ICF.
15. Being pregnant or breast feeding, or planning to become pregnant or give birth during this trial.
16. Having received any live attenuated vaccine within 4 weeks prior to investigational product or planning to receive such vaccines during the study.
17. Having undergone a major surgery.
18. Any diseases that at the investigator's discretion may confound the trial results, interfere with the participation in the entire trial, and/or would make participating in the trial not in the participant's best interest, or a medical history with treatment or laboratory abnormalities, or any other circumstances that would make it inappropriate for the participant to be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate in patients with CIS | 3,6,12 months time point from the date of the first dose of T3011
Recurrence Free Survival Rate in patients with Ta/T1 (without CIS) | 3,6,12 months time point from the date of the first dose of T3011
Incidence rates of Grade ≥3 treatment-related adverse events (TRAEs) | 24 months
Incidence rates of TRAEs leading to treatment discontinuation, dose modification or treatment interruption. | 24 months

SECONDARY OUTCOMES:
Complete Response Rate in patients with CIS | 18,24 months time point from the date of the first dose of T3011
Recurrence Free Survival Rate in patients with Ta/T1 (without CIS) | 18,24 months time point from the date of the first dose of T3011
Safety Endpoints | 24 months
  * Incidence rates of Grade ≥3 treatment-emergent adverse events (TEAEs)
  * Incidence rates of all grades of TRAEs
  * Incidence rates of AEs leading to treatment discontinuation, dose modification or treatment interruption

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - East Valley Urology Center, Queen Creek, Arizona
  - Florida Urology Partners, LLP, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No